CLINICAL TRIAL: NCT06619457
Title: Evaluation of the Anti-aging Efficacy of One Face Care Cosmetic Product
Acronym: SkinBioAge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amazentis SA (Industry)
Collaborators: proDERM GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 24.0199-23
Record Dates: First submitted 2024-09-25; First posted 2024-10-01 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2024-10

CONDITIONS: Skin Aging
Keywords: Mitochondria; Urolithin A; Mitopure; Aging
MeSH Terms: interventions — 3,8-dihydroxy-6H-dibenzo(b,d)pyran-6-one

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo Cream (Experimental)
  Interventions: Other: Placebo Cream
- Active Moisturizing Cream (Experimental)
  Interventions: Other: Mitopure (Urolithin A) Cream

INTERVENTIONS:
Other: Mitopure (Urolithin A) Cream — cosmetic cream to be applied topically on face and forearms twice/daily using split/face design
  Arms: Active Moisturizing Cream
Other: Placebo Cream — cosmetic cream to be applied topically on face and forearms twice/daily using split/face design
  Arms: Placebo Cream

SUMMARY:
The purpose of this study is to evaluate the anti-wrinkle efficacy and effect on skin epigenetic and on mitochondrial morphology of a facial cosmetic product compared to a placebo

ELIGIBILITY:
Inclusion Criteria:

* Written Informed Consent to participate in the study
* Willingness to actively participate in the study and to come to the scheduled visits
* Female and approximately 10% male (at least 4 male subjects)
* From 50 to 75 years of age
* Healthy skin in the test areas
* Visible wrinkles in the face (grade 3 to 6 according to SGS proderm scale)

For biopsy subpanel:

-Vaccination of tetanus within the last 10 years

Exclusion Criteria:

* Female subjects: Pregnancy or lactation
* Drug addicts, alcoholics
* AIDS, HIV-positive or infectious hepatitis
* Conditions which exclude a participation or might influence the test reaction/evaluation
* Participation or being in the waiting period after participation in cosmetic and/or pharmaceutical studies pertaining to the test area
* Active skin disease at the test area
* Documented allergies to face/eye care products
* Diabetes mellitus
* Cancer not being diagnosed as cured and requiring chemotherapy, irradiation and/or hormonal treatment within the last 2 years
* One of the following illnesses with reduced physical capability/fitness: asthma (symptom-free allergic asthma is not an exclusion criterion), hypertension (if not adjusted with medication), cardiovascular diseases
* Epilepsy
* Wounds, moles, tattoos, scars, irritated skin, excessive hair growth, freckles, etc. at the test area that could influence the investigation
* Regular use of tanning beds
* Any topical medication at the test area within the last 3 days prior to the start of the study
* Systemic therapy with immuno-suppressive drugs (e.g. corticosteroids) and/or antihistamines (e.g. antiallergics) and/or within the last 7 days prior to the start of the study
* Therapy with antibiotics within the last 2 weeks prior to the start of the study
* Past cosmetic surgery procedure in the test area (e.g. laser, facelift)
* Cosmetic surgery procedure in the test area, e.g. IPL (Intensed Pulsed Light), botox, chemical peel, dermabrasion within the last 2 years prior to the start of the study and/or throughout the entire course of the study
* Medical treatment for wrinkle reduction (e.g. peeling with vitamin A or fruit acids) on the face within the last 2 weeks prior to the start of the study

For biopsy subpanel:

* Regular medication with anti-coagulating drugs like Aspirin®, Macumar®, etc. (e.g. for thrombosis prophylaxis) within up to 15 days prior to the taking of the biopsies
* History of complications at wound healing (e.g. keloids, hypertrophic scars or contracture scar)
* Known intolerance to local anaesthetics
* Known Sensitivity to any dressing systems

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2024-09-25 (Actual); Primary Completion 2024-12-12 (Actual); Study Completion 2024-12-12 (Actual)

PRIMARY OUTCOMES:
Anti-wrinkle efficacy | 12 weeks
  Anti-wrinkle efficacy will be assessed in the periorbital regions wrinkles using AEVA. Parameters measured: Rz and Ra, representing mainly the rough structure (Rz) or the finer skin structure (Ra).
Skin Biological age | 12-weeks
  DNA methylation patterns analysis (epigenetics) by skin tape stripping (D-Squames)

SECONDARY OUTCOMES:
Skin hydration | 12 weeks
  Change from baseline in skin hydration (assessed on skin capacitance by Corneometer [a.u.])
Transepidermal Water Loss (TEWL) | 12 weeks
  Change from baseline in skin barrier function (assessed as transepidermal waterloss by Tewameter [g/(m²h)])
Mitochondrial morphology in skin | 12 weeks
  mitochondrial morphology in skin will be assessed via transmission electron microscopy (TEM) on 3mm punch-biopsies
Photodocumentation of skin health | 12 weeks
  ColorFace image analysis of face via facial photography
Subjective questionnaire | 12 weeks
  Subjective evaluation of product traits assessed via questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Katrin Unbereit, PhD, Principal Investigator — SGS proderm GmbH
Locations (1):
- SGS proderm GmbH, Schenefeld, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No